CLINICAL TRIAL: NCT05244096
Title: A Retrospective Chart Review Study to Determine the Effects of Psychotropic Medications and Prior Psychiatric Diagnoses on COVID-19 Patients' Disease Progression, and Severity.
Brief Title: COVID-19 & Psychiatry: A Retrospective Chart Review
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jeffrey Rado, Associate Professor, Northwestern University
Other Study IDs: STU00214993
Record Dates: First submitted 2022-02-15; First posted 2022-02-17 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID+: COVID + positive individuals from March 15 2020 to Nov 30, 2021
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study

SUMMARY:
A retrospective chart review study to determine the effects of psychotropic medications and prior psychiatric diagnoses on COVID-19 patients' disease progression, and severity.

DETAILED DESCRIPTION:
The goal of this study would be to study the association between use of psychotropic medications and prior psychiatric diagnoses on COVID-19 patients' disease progression and severity.

ELIGIBILITY:
Inclusion Criteria:

- Individuals with a positive COVID-19 test between March 15 2020 to November 30 2021 at Northwestern Medicine hospitals.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19
Sampling Method: Probability Sample
Enrollment: 65000 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Hazard Ratio | March 15 2020 to Nov 30 2021
  HR of using psych drugs or having psych diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rado, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwester Clinical Research Program, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No